CLINICAL TRIAL: NCT02903940
Title: The Application of Negative Atrioventricular Hysteresis in Cardiac Resynchronization Therapy
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD_855
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CRT+NAVH: Surface ECG recordings will be taken during the adjustment of programmable Cardiac Resynchronization Therapy and Negative Atrioventricular Hysteresis settings.
  Interventions: Device: CRT+NAVH

INTERVENTIONS:
Device: CRT+NAVH — Cardiac Resynchronization Therapy with Negative Atrioventricular Hysteresis

SUMMARY:
The purpose of this study is to evaluate the application of Negative Atrioventricular Hysteresis (NAVH) to improve electrical synchrony in Cardiac Resynchronization Therapy (CRT) patients.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a functioning SJM Quadripolar CRT Pacing System
* QRS duration > 140 ms
* Left bundle branch block documented
* Ability to provide informed consent for study participation
* Willing to comply with the study evaluation requirements
* At least 18 years of age

Exclusion Criteria:

* CRT Pacing System implanted less than 1 week at time of enrollment
* CRT Pacing System implanted more than 24 months at time of enrollment
* CRT Pacing System implanted more than 90 days at time of enrollment AND intrinsic QRS duration is shorter than pre-implant intrinsic QRS duration by more than 10 ms
* Resting ventricular rate >100 bpm
* Intrinsic PR interval > 300 ms
* Paroxysmal or persistent atrial tachycardia or atrial fibrillation documented
* A recent myocardial infarction, ablation, drug intoxication, electrolyte imbalance, or any condition within the last 90 days that would be contraindicated for CRT programming changes in the opinion of the investigator
* Women who are pregnant or who plan to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already implanted with SJM Quadripolar CRT Pacing Systems will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Acute changes in surface ECG QRS duration resulting from Cardiac Resynchronization Therapy with Negative Atrioventricular Hysteresis over a range of programmable values | 1 day

SECONDARY OUTCOMES:
Ambulatory changes in surface ECG QRS duration resulting from Cardiac Resynchronization Therapy with Negative Atrioventricular Hysteresis | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No